CLINICAL TRIAL: NCT02481778
Title: Monitoring Radiation Induced Cardiac Damage by Blood Markers
Acronym: CARD
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: RT2014-01
Record Dates: First submitted 2015-05-11; First posted 2015-06-25 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Radiation Induced Cardiac Damage
Keywords: Radiotherapy; Cardiac; Toxicity
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood sampling

SUMMARY:
Rationale:

Radiation induced cardiac toxicity after treatment for intrathoracic tumours is a clinically relevant problem. So far, no clinical prediction models exist for cardiac toxicity. In particular, the relationship between radiation dose parameters and the risk of cardiac toxicity remains to be determined.

Clinical prediction models for cardiac toxicity are difficult to obtain, e.g. due to long latency time. Therefore, objective surrogate markers, for cardiac toxicity such as NT pro BNP and hs-TNT, as obtained during and after treatment may be of great value.

Objective:

The main objective to find a correlation between the rise in NT pro BNP level and the radiation dose given to the heart.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven oesophageal- or lung cancer (adeno-, or squamous cell carcinoma or other NSCLC type)
* Older than 18 years
* Written informed consent

Exclusion Criteria:

* Prior radiotherapy to the chest including radiotherapy for breast cancer
* Patients treated with palliative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal- or non small cell lung cancer treated with radiotherapy with curative intention, with or without chemotherapy, with or without surgery, at the department of radiotherapy at the University Medical Centre Groningen
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Change in percentage of rise of the level of NT pro BNP after radiotherapy | At 1 year after end of radiation therapy

SECONDARY OUTCOMES:
Cardiac events | After start treatment up to 2 years after end of radiation therapy.
  A new diagnosis of: heart failure, myocardial infarction or a newly diagnosed rhythm disorder will be scored as a cardiac event. Myocardial ischaemia requiring intervention and changes in cardiac medication in case of deterioration of known heart failure will be analysed by a cardiologist to decide whether or not to score this as an event. Events will be scored according the CTCAE 4.2 criteria.
Change in percentage of rise of hs-TNT during or after treatment | At day 1 start radiation therapy and at last day of radiation therapy (an expected average of 5 weeks after start of radiation therapy) and at 4 weeks, 6 months, 1 and 2 years after end of radiation therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands